CLINICAL TRIAL: NCT02170363
Title: HeartMate 3™ CE Mark Clinical Investigation Plan
Acronym: HM3 CE Mark
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Center for Life Sciences (Unknown); Emergo (Unknown); KCRI (Other); Thoratec Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TC02212014
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Advanced Refractory Left Ventricular Heart Failure
Keywords: Heart Failure; Ventricular Dysfunction; Cardiomyopathies; Heart Disease; Cardiovascular Disease; Heart-assist devices; Thoratec Corporation
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction; Cardiomyopathies; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HeartMate 3 (Experimental): Left Ventricular Assist System (LVAS) to be used on Subjects with advanced refractory left ventricular heart failure
  Interventions: Device: Left Ventricular Assist System (LVAS)

INTERVENTIONS:
Device: Left Ventricular Assist System (LVAS) — Implantation of left ventricular assist device for hemodynamic support

SUMMARY:
The purpose of this clinical investigation is to evaluate the performance and safety of the HeartMate 3 Left Ventricular Assist System (HM3 LVAS) To support obtaining CE Mark for the HM3 LVAS in Europe, a multi-center clinical study will be conducted in multiple countries. The clinical study will be conducted in compliance with the Declaration of Helsinki, ICH/GCP and EN ISO 14155:2011 Requirements for Clinical Investigations and in accordance with country-specific requirements, under one clinical study protocol.

This study will evaluate the performance of the HM3 LVAS, side effects and undesirable conditions within acceptable risks and weigh them against the intended performance of HM3 LVAS in accordance with Essential Requirements 2, 5 and 16 of the Active Implantable Medical Device Directive 90/385/EEC (AIMDD).

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legal representative has signed Informed Consent Form (ICF)
2. Age ≥ 18 years
3. BSA ≥ 1.2 m2
4. NYHA IIIB or IV OR ACC/AHA Stage D
5. LVEF ≤ 25%
6. CI ≤ 2.2 L/min/m2, while not on inotropes
7. Patients must also meet one of the following:

   - On Optimal Medical Management (OMM), based on current heart failure practice guidelines for at least 45 out of the last 60 days and are failing to respond,

   OR

   - In NYHA class IIIB or IV heart failure for at least 14 days AND dependent on intraaortic balloon pump (IABP) for at least 7 days,

   OR

   - Inotrope dependent/unable to wean from inotropes

   OR

   - Listed for Transplant
8. Females of child bearing age must agree to use adequate contraception

Exclusion Criteria:

1. Etiology of HF due to or associated with uncorrected thyroid disease, obstructive cardiomyopathy, pericardial disease, amyloidosis or restrictive cardiomyopathy
2. Technical obstacles which pose an inordinately high surgical risk, in the judgment of the investigator
3. Existence of ongoing mechanical circulatory support (MCS) other than IABP
4. Positive pregnancy test if of childbearing potential
5. Lactating mothers
6. Presence of mechanical aortic cardiac valve that will not be converted to a bioprosthesis at the time of LVAD implant
7. History of any organ transplant
8. Platelet count < 100,000 x 103/L (< 100,000/ml)
9. Psychiatric disease/disorder, irreversible cognitive dysfunction or psychosocial issues that are likely to impair compliance with the study protocol and LVAS management
10. History of confirmed, untreated AAA > 5 cm in diameter
11. Presence of an active, uncontrolled infection
12. Intolerance to anticoagulant or antiplatelet therapies or any other peri/post-operative therapy the investigator will require based upon the patients' health status
13. Presence of any one of the following risk factors for indications of severe end organ dysfunction or failure:

    1. An INR ≥ 2.5 not due to anticoagulation therapy
    2. Total bilirubin > 43 umol/L (2.5 mg/dl), shock liver, or biopsy proven liver cirrhosis
    3. History of severe chronic obstructive pulmonary disease (COPD) defined by FEV1/FVC < 0.7, or FEV1 <50% predicted
    4. Fixed pulmonary hypertension with a most recent PVR ≥ 8 Wood units that is unresponsive to pharmacologic intervention
    5. History of stroke within 90 days prior to enrollment, or a history of cerebrovascular disease with significant (> 80%) carotid artery stenosis
    6. Serum creatinine ≥221umol/L (2.5 mg/dl) or the need for chronic renal replacement therapy
    7. Significant peripheral vascular disease (PVD) accompanied by rest pain or extremity ulceration
14. Patient has moderate to severe aortic insufficiency without plans for correction during pump implant
15. Pre albumin < 150 mg/L, or Albumin < 30g/L (3 g/dL)
16. Planned Bi-VAD support prior to enrollment
17. Patient has known hypo or hyper coagulable states such as disseminated intravascular coagulation and heparin induced thrombocytopenia
18. Participation in any other clinical investigation that is likely to confound study results or affect the study
19. Any condition other than HF that could limit survival to less than 24 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2020-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Gazzola, B. Sc., Study Director — Abbott
Locations (10):
- The Alfred Hospital, Melbourne, Victoria, Australia
- AKH Medical University of Vienna, Vienna, Austria
- Toronto General Hospital, Toronto, Ontario, Canada
- Institute for Clinical and Experimental Medicine (IKEM), Prague, Czechia
- Germany (5):
  - Herz- und Diabeteszentrum NRW Thorax- und Kardiovaskularchirurgie Clinic, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - Universitats-Herzzentrum Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Herzentrum Leipzig GmbH, Leipzig
- National Research Center for Cardiac Surgery, Astana, Kazakhstan

REFERENCES:
- [Result] Netuka I, Sood P, Pya Y, Zimpfer D, Krabatsch T, Garbade J, Rao V, Morshuis M, Marasco S, Beyersdorf F, Damme L, Schmitto JD. Fully Magnetically Levitated Left Ventricular Assist System for Treating Advanced HF: A Multicenter Study. J Am Coll Cardiol. 2015 Dec 15;66(23):2579-2589. doi: 10.1016/j.jacc.2015.09.083. PMID 26670056
- [Derived] Schmitto JD, Pya Y, Zimpfer D, Krabatsch T, Garbade J, Rao V, Morshuis M, Beyersdorf F, Marasco S, Sood P, Damme L, Netuka I. Long-term evaluation of a fully magnetically levitated circulatory support device for advanced heart failure-two-year results from the HeartMate 3 CE Mark Study. Eur J Heart Fail. 2019 Jan;21(1):90-97. doi: 10.1002/ejhf.1284. Epub 2018 Jul 27. PMID 30052304
- [Derived] Krabatsch T, Netuka I, Schmitto JD, Zimpfer D, Garbade J, Rao V, Morshuis M, Beyersdorf F, Marasco S, Damme L, Pya Y. Heartmate 3 fully magnetically levitated left ventricular assist device for the treatment of advanced heart failure -1 year results from the Ce mark trial. J Cardiothorac Surg. 2017 Apr 4;12(1):23. doi: 10.1186/s13019-017-0587-3. PMID 28376837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 50 patients were recruited at 10 cardiac transplant centers and implanted between June 25, 2014, and November 27, 2014
Pre-assignment Details: The data presented in this record includes all 50 patients followed through to the 6-month primary endpoint.
Groups:
- HeartMate 3: HeartMate 3 Left Ventricular Assist System (HM3 LVAS) used for advanced refractory left ventricular heart failure (50 Subjects in the Study Cohort).
Period: Overall Study
Arm/Group | HeartMate 3
Started | 50
Completed | 50 (Followed to the 6-Month Primary Endpoint)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HeartMate 3
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.9 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 45
Region of Enrollment [Number; unit: participants]
  Canada | 3
  Austria | 7
  Czech Republic | 10
  Australia | 1
  Kazakhstan | 8
  Germany | 21
Body Surface Area [Mean (Standard Deviation); unit: M^2] — Body Surface Area (BSA) calculated from patients height and weight
  M^2 | 2 (0.2)
Cardiac Index [Mean (Standard Deviation); unit: L/min/m^2] — Cardiac index (CI) is a hemodynamic parameter that relates the cardiac output (CO) from left ventricle in one minute to body surface area (BSA), thus relating heart performance to the size of the individual. Values less than 2.2 L/min/m^2 indicate that the patient may be in cardiogenic shock.
  L/min/m^2 | 1.8 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Comparison of survival at 6 months of Left Ventricular Assist Device (LVAD) support to a performance goal established using matched HeartMate II INTERMACS data
Time Frame: 6 months
Population: All 50 patients were analyzed when the last patient reached the 6-month primary endpoint on May 26, 2015
Measure: Number (97.5% Confidence Interval); unit: Percentage of Participants who Survived
Arm/Group | HeartMate 3
Number analyzed (Participants) | 50
Percentage of Participants who Survived | 92 [83 to 97]

2. Secondary Outcome: Quality of Life (EQ-5D-5L)
Description: The EQ-5D-5L is a standardized measure of health status developed by the EuroQol Group. Patients describe their perceived health status using an analog scale with 0 as the worst health the patient can imagine and 100 as the best health (Visual Analog Score). The patients' scores at one, three and six months were compared to their baseline scores and the resulting positive scores indicated improved quality of life.
Time Frame: Baseline, Month 1, Month 3, Month 6
Population: Patients alive and capable of performing the test at 6 months
Measure: Median (Full Range); unit: Units on a EQ-5D-5L Score scale
Arm/Group | HeartMate 3
Number analyzed (Participants) | 50
Units on a EQ-5D-5L Score scale
  Baseline: number analyzed (Participants) | 43
  Baseline | 50 [12 to 90]
  Month 1: number analyzed (Participants) | 43
  Month 1 | 60 [10 to 95]
  Month 3: number analyzed (Participants) | 43
  Month 3 | 70 [30 to 100]
  Month 6: number analyzed (Participants) | 40
  Month 6 | 75 [29 to 100]

3. Secondary Outcome: Functional Status - Six Minute Walk Test (6MWT)
Description: The Six Minute Walk Test(6MWT)measures the distance that a patient can walk in a period of 6 minutes. The distance walked is measured in meters. This test measures the patients' functional status. The more meters a patient can walk over baseline indicates improvement in functional status.
Time Frame: Baseline, Month 1, Month 3, Month 6
Population: Only patients alive, capable and willing to perform test are included.
Measure: Median (Full Range); unit: meters
Arm/Group | HeartMate 3
Number analyzed (Participants) | 50
meters
  Baseline | 236 [5 to 550]
  Month 1: number analyzed (Participants) | 49
  Month 1 | 260 [21.1 to 582]
  Month 3: number analyzed (Participants) | 47
  Month 3 | 375 [35 to 671]
  Month 6: number analyzed (Participants) | 44
  Month 6 | 385 [70 to 705]

4. Secondary Outcome: Functional Status - New York Heart Association (NYHA) Classification
Description: NYHA classification relates symptoms to every day activities and patients quality of life. Class 1 = no limitations on physical activity Class 2 - slight limitation of physical activity Class 3 - marked limitation of physical activity Class 4 = unable to carry out any physical activity without discomfort
Time Frame: Baseline, Month 1, Month 3, Month 6
Population: Only patients alive, capable and willing to perform test are included.
Measure: Number; unit: percentage of participants
Arm/Group | HeartMate 3
Number analyzed (Participants) | 50
percentage of participants
  Baseline NYHA I or II | 0
  Baseline NYHA III or IV | 100
  Month 1 NYHA I or II: number analyzed (Participants) | 44
  Month 1 NYHA I or II | 64
  Month 1 NYHA III or IV: number analyzed (Participants) | 44
  Month 1 NYHA III or IV | 36
  Month 3 NYHA 1 or II: number analyzed (Participants) | 43
  Month 3 NYHA 1 or II | 81
  Month 3 NYHA III or IV: number analyzed (Participants) | 43
  Month 3 NYHA III or IV | 19
  Month 6 NYHA I or II: number analyzed (Participants) | 42
  Month 6 NYHA I or II | 83
  Month 6 NYHA III or IV: number analyzed (Participants) | 42
  Month 6 NYHA III or IV | 17

5. Secondary Outcome: All Adverse Events
Description: Frequency of pre-defined anticipated adverse events
Time Frame: As they occurred, Baseline through 180 Days
Measure: Number; unit: % of Participants with Adverse Events
Arm/Group | HeartMate 3
Number analyzed (Participants) | 50
% of Participants with Adverse Events
  Bleeding | 38
  Bleeding requiring surgery | 14
  Gastrointestinal bleeding | 8
  Cardiac Arrhythmia | 34
  Pericardial fluid | 2
  Internal device malfunction | 6
  Pump thrombosis | 0
  External device malfunctions | 24
  Hemolysis | 0
  Hepatic dysfunction | 2
  Hypertension | 2
  Any infection | 36
  Infection - sepsis | 16
  Infection - driveline | 10
  Myocardial infarction | 0
  Any stroke | 12
  Stroke - ischemic | 8
  Stroke - hemorrhagic | 4
  Neurologic dysfunction | 8
  Psychiatric episode | 6
  Renal dysfunction | 10
  Respiratory failure | 16
  Right heart failure | 10
  Right heart failure w RVAD | 4
  Wound dehiscence | 8
  Other | 54

6. Secondary Outcome: Device Malfunctions
Description: Frequency and incidence of device malfunction
Time Frame: As they occurred, Baseline through 180 Days; Subjects that remain ongoing after 6 months will continue to be followed to 24 months post-implant or outcome
Measure: Number; unit: Number of events
Arm/Group | HeartMate 3
Number analyzed (Participants) | 50
Number of events
  Pump malfunctions | 0
  Non-pump malfunction: internal component | 3
  Non-pump malfunction: External components | 14

7. Secondary Outcome: Reoperations
Description: Frequency of reoperations
Time Frame: As they occurred, Baseline through 180 Days
Population: Twenty-nine (58%) did not have reoperation
Measure: Number; unit: Number of re-operations by reason
Arm/Group | HeartMate 3
Number analyzed (Participants) | 50
Number of re-operations by reason
  Major bleeding | 11
  Cardiac arrhythmia | 1
  Pericardial fluid | 1
  Major infection | 3
  Respiratory failure | 4
  Right heart failure | 3
  Wound dehiscence | 15
  Other | 23

8. Secondary Outcome: Rehospitalizations
Description: Frequency and incidence of rehospitalizations
Time Frame: As they occurred, Baseline through 180 Days
Population: Number of Participants with Rehospitalizations According to Rehospitalization Type
Measure: Count of Participants; unit: Participants
Arm/Group | HeartMate 3
Number analyzed (Participants) | 43
Participants
  Suspected device malfunction | 1
  Transplant/ Transplant evaluation | 1
  Anticoagulation maintenance | 1
  Routine testing | 1
  ICD therapy | 1
  Suspected driveline infection | 1
  Bleeding | 4
  Infection | 6
  Neurologic dysfunction | 1
  Arrythmia | 1
  Volume issue | 3
  INR | 5
  Chest pain | 2
  Other | 9

9. Secondary Outcome: Stroke Free Survival
Description: Percentage of participants free of debilitating stroke (Modified Rankin Score > 3)
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | HeartMate 3
Number analyzed (Participants) | 50
percentage of participants | 90

ADVERSE EVENTS:
Time Frame: From time of device implant to 6 months
Description: Adverse events were documented by study site staff as they occurred per protocol definitions.
Arm/Group | HeartMate 3
All-Cause Mortality (participants affected / at risk) | 4/50
Serious Adverse Events (participants affected / at risk) | 34/50
Other Adverse Events (participants affected / at risk) | 34/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HeartMate 3 (N=50)
Bleeding (General disorders) | 14 (19)
Bleeding - Requiring Surgery (Blood and lymphatic system disorders) | 7 (8)
Bleeding - Gastrointestinal (Blood and lymphatic system disorders) | 4 (6)
Cardiac Arrhythmias - Ventricular (Cardiac disorders) | 6 (6)
Cardiac Arrhythmias - Supraventricular (Cardiac disorders) | 0 (0)
Pericardial Fluid (Cardiac disorders) | 1 (1)
Internal Device Malfunction (Surgical and medical procedures) | 1 (1)
Pump Thrombosis (Product Issues) | 0 (0)
External Device Malfunctions (Product Issues) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 0 (0)
Hepatic Dysfunction (Hepatobiliary disorders) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0)
Any Infection (Infections and infestations) | 11 (13)
Infection - Sepsis (Infections and infestations) | 6 (6)
Infection - Driveline (Infections and infestations) | 3 (3)
Infection - Pump (Infections and infestations) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0)
Any Stroke (Nervous system disorders) | 6 (6)
Stroke - Ischemic (Nervous system disorders) | 4 (4)
Stroke - Hemorrhagic (Nervous system disorders) | 2 (2)
Neurologic Dysfunction (Nervous system disorders) | 1 (1)
Psychiatric Episode (Psychiatric disorders) | 1 (1)
Renal Dysfunction (Renal and urinary disorders) | 3 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Right Heart Failure (Cardiac disorders) | 4 (4)
Right Heart Failure - requiring RVAD (Cardiac disorders) | 2 (2)
Arterial Thromboembolism (Blood and lymphatic system disorders) | 0 (0)
Venous Thromboembolism (Blood and lymphatic system disorders) | 0 (0)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 3 (3)
Other Serious Adverse Event (General disorders) | 17 (24)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HeartMate 3 (N=50)
Bleeding (Blood and lymphatic system disorders) | 5 (16)
Cardiac Arrhythmias (Cardiac disorders) | 11 (11)
Cardiac Arrhythmias - Supraventricular (Cardiac disorders) | 10 (10)
External Device Malfunction (Product Issues) | 11 (13)
Any infection (Infections and infestations) | 7 (15)
Neurologic Dysfunction (Nervous system disorders) | 3 (3)
Other Non-serious Adverse Event (General disorders) | 10 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days